CLINICAL TRIAL: NCT05098769
Title: A Predictive Tool for Predicting Adverse Outcomes in Acute Pulmonary Embolism Patients Using Parameters Obtained by Computed Tomographic Pulmonary Angiography.
Brief Title: A Predictive Tool for Predicting Adverse Outcomes in Acute Pulmonary Embolism Patients Using CTPA.
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, YIZHUO GAO, Principal Investigator, Shengjing Hospital
Other Study IDs: AOAPECT
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Embolism and Thrombosis; Deterioration, Clinical
Keywords: Pulmonary Embolism and Thrombosis; Deterioration, Clinical
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis; Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute pulmonary embolism: an age of ≥ 18 years and a PE diagnosis based on CT pulmonary angiography

SUMMARY:
This study collected clinical, laboratory, and CT parameters of acute patients with acute pulmonary embolism from admission to predict adverse outcomes within 30 days after admission into hospital.

DETAILED DESCRIPTION:
This study collected clinical, laboratory, and CT parameters of acute patients with acute pulmonary embolism from admission. The outcomes of interest were defined as the occurrence of adverse outcomes within 30 days after admission into hospital.

Eligible patients were randomized in some ratio into derivation and validation cohorts. The derivation cohort was used to develop and evaluate a multivariable logistic regression model for predicting the outcomes of interest. The discriminatory power was evaluated by comparing the nomogram to the established risk stratification systems. The consistency of the nomogram was evaluated using the validation cohort.

ELIGIBILITY:
Inclusion Criteria:

* age of ≥ 18 years and a PE diagnosis based on CT pulmonary angiography

Exclusion Criteria:

* pregnancy
* reception of reperfusion treatment before admission
* missing data regarding CT parameters, echocardiography, cardiac troponin I (c-Tn I), and N-terminal-pro brain natriuretic peptide (NT-pro BNP) levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse outcomes | 30 days
  The outcomes of interest were defined as the occurrence of adverse outcomes within 30 days after admission. Adverse outcomes were defined as PE-related deaths, the need for mechanical ventilation, the need for cardiopulmonary resuscitation, and the need for life-saving vasopressor and reperfusion treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenjing Hospital of CHINA MEDICAL UNIVERSITY, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Gao Y, Gu Z, Wei X, Wei S, Liu Y, Zhan S, Yang J, Qi C, Qi S, Wang M, Jia D. Ventricular septum curvature ratio: a novel imaging marker to predict clinical deterioration in normotensive acute pulmonary embolism. Crit Care. 2025 Oct 31;29(1):463. doi: 10.1186/s13054-025-05708-w. PMID 41174707
- [Derived] Gao Y, Wei S, Liu Y, Yu Z, Zhan S, Yang B, Qi C, Qi S, Wang M, Jia D. Predicting Deterioration in Patients With Normotensive Acute Pulmonary Embolism Using Clinical-Imaging Features: A Multicenter Prospective Cohort Study. J Am Heart Assoc. 2025 Jul;14(13):e038984. doi: 10.1161/JAHA.124.038984. Epub 2025 Jun 27. PMID 40576035